CLINICAL TRIAL: NCT03628300
Title: Neurotoxicity Evaluation of Beta-lactams in Intensive Care Unit and Identification of the Risk Factors
Acronym: NebuLar
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0036
Record Dates: First submitted 2018-07-30; First posted 2018-08-14 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2018-08

CONDITIONS: Neurotoxicity; Sepsis; Beta Lactams; Therapeutic Drug Monitoring; Critical Care; Acute Kidney Injury
Keywords: neurotoxicity; Sepsis; beta lactams; therapeutic drug monitoring; critical care; Acute Kidney Injury
MeSH Terms: conditions — Neurotoxicity Syndromes; Sepsis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Beta-lactams are the most prescribed antibiotics in intensive care units. The lack of linearity between the dose administered and the exposition due to the very high variability of the pharmacokinetics in critically ill patients requires that the treatment be adapted on a case-by-case basis depending on the drug serum concentration. However, maximum concentrations not to be exceeded in order to limit beta-lactams toxicity are generally unknown. The main toxic risk of beta-lactams in intensive care is indeed neurological, but the neurotoxicity is probably underdiagnosed due to the variability of the signs observed, their time to onset, and confounding factors. Apart from recommendations for dose adjustment in the event of renal insufficiency, the procedures for the proper use of beta-lactams in intensive care are poorly established. The study presented here aims to assess the impact of the neurotoxic risk of beta-lactams in intensive care based on therapeutic drug monitoring, and thus to improve beta-lactam safety in critically ill patients.

This is a prospective cohort study evaluating change in neurological status of patients admitted to the ICU and treated with a beta-lactam antibiotic with therapeutic drug monitoring. Neurological evaluation and scoring (Glasgow scale, CAM-ICU, Richmond agitation-sedation scale) and beta-lactam serum concentration assay are performed together 2 to 3 times a week.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU
* Treatment initiation by an antibiotic of the beta-lactam class
* Beta-lactam therapeutic drug monitoring

Exclusion criteria:

* Any neurological disorder already present at admission
* Patients on mechanical ventilation who presented a neurological disorder before being intubated and sedated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective cohort study evaluating change in neurological status of patients admitted to the ICU and treated with a beta-lactam antibiotic with therapeutic drug monitoring. Neurological evaluation and scoring (Glasgow scale, CAM-ICU, Richmond agitation-sedation scale) and beta-lactam serum concentration assay are performed together 2 to 3 times a week.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
proportion of patients with a change in neurological status | one week
  the primary objective is to assess the frequency of beta-lactam neurotoxicity in a standardized use with therapeutic drug monitoring

SECONDARY OUTCOMES:
beta-lactam serum concentration according neurological status | one week
  beta-lactam serum concentration is assayed by a validated HPLC method

CONTACTS AND LOCATIONS:
Overall Officials: Youssef Youssef, MD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No